CLINICAL TRIAL: NCT03864926
Title: Envarsus in Delayed Graft Function: A Phase IV, Randomized, Single Center Study Among Kidney Transplant Recipients With Delayed Graft Function (DGF) to Study the Effect of Envarsus XR in the DGF Recovery
Brief Title: Envarsus in Delayed Graft Function (E-DGF)
Acronym: E-DGF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0530; A534280 (Other: UW Madison); SMPH/MEDICINE/NEPHROLOGY (Other: UW Madison)
Record Dates: First submitted 2019-03-05; First posted 2019-03-06 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-05

CONDITIONS: Delayed Graft Function
Keywords: Kidney Transplant
MeSH Terms: conditions — Delayed Graft Function | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (Active Comparator): Standard of Care Tacrolimus
  Interventions: Drug: Tacrolimus
- Experimental (Experimental): Envarsus XR
  Interventions: Drug: Envarsus XR

INTERVENTIONS:
Drug: Envarsus XR — Envarsus XR is FDA approved for the prophylaxis of organ rejection in kidney transplant recipients converted from tacrolimus immediate-release formulations, in combination with other immunosuppressants. Envarsus XR, is designed to deliver tacrolimus more smoothly over the whole day.
  Envarsus XR, a calcineurin-inhibitor immunosuppressant, is available for oral administration as extended-release tablets containing the equivalent of 0.75 mg, 1 mg, or 4 mg of anhydrous tacrolimus USP. Inactive ingredients include hypromellose USP, lactose monohydrate NF, polyethylene glycol NF, poloxamer NF, magnesium stearate NF, tartaric acid NF, butylated hydroxytoluene NF, and dimethicone NF. Tacrolimus is the active ingredient in ENVARSUS XR.
  Arms: Experimental
Drug: Tacrolimus — Tacrolimus (generic; immediate release) is FDA approved for the prophylaxis of organ rejection in heart, kidney and liver transplant recipients.
  Arms: Standard of Care

SUMMARY:
Envarsus XR is an extended release tacrolimus designed to deliver tacrolimus more consistently, thus avoiding large fluctuations of tacrolimus trough levels with Envarsus XR compared to immediate release tacrolimus. It is expected that patients with DGF on Envarsus XR will have more stable tacrolimus levels and facilitate early recover from DGF compared to immediate release tacrolimus.

DETAILED DESCRIPTION:
This is a single center randomized phase IV trial of comparing extended release Envarsus XR (study drug) once a day vs immediate release tacrolimus twice a day in a new kidney transplant recipients with delayed graft function (DGF). The primary study endpoint is the interval between first dialysis and last dialysis after kidney transplant (duration of DGF). The second end point is the number of tacrolimus or Envarsus XR dose adjustments required during the period of DGF.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Willing to comply with all study procedures and be available for the duration of the study
3. Male or female, at least 18 years of age
4. Documented diagnosis of DGF or need for dialysis or had dialysis within the first week of kidney transplant
5. Current treatment with tacrolimus based regimen or planned to start tacrolimus based immunosuppressive regimen
6. Females of childbearing potential must have a negative urine or serum pregnancy test prior to randomization and agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to randomization, for the duration of study participation, and for 7 days following completion of therapy.

   * A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

     * Has not undergone a hysterectomy or bilateral oophorectomy; or
     * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

1. History of hypersensitivity or allergy to any of the study drugs or drugs of similar chemical classes
2. Current use of non-tacrolimus based immunosuppressive regimen or no plan to start tacrolimus based regimen
3. Women who are or plan to become pregnant or breast-feeding during the study period
4. Not suitable for study participation due to other reasons at the discretion of the investigator
5. Major post-surgical complications requiring allograft nephrectomy
6. Multi-organ transplant recipients
7. Non kidney transplant recipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandesh Parajuli, MBBS, Principal Investigator — University of Wisconsin School of Medicine and Public Health, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Parajuli S, Bloom M, Mandelbrot D, Astor BC. Serum beta2-Microglobulin Predicts Time to Recovery of Delayed Graft Function in Kidney Transplant Recipients. Clin Transplant. 2024 Aug;38(8):e15435. doi: 10.1111/ctr.15435. PMID 39158946

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the University of Wisconsin Hospital and Clinics between March 2019 and April 2022.
Groups:
- Standard of Care: Tacrolimus (generic; immediate release) is FDA approved for the prophylaxis of organ rejection in heart, kidney and liver transplant recipients.
  Dosage was clinically determined, dose form was oral tablets, and SOC tacrolimus was twice daily
- Experimental: Envarsus XR is FDA approved for the prophylaxis of organ rejection in kidney transplant recipients converted from tacrolimus immediate-release formulations, in combination with other immunosuppressants. Envarsus XR, is designed to deliver tacrolimus more smoothly over the whole day.
  Envarsus XR, a calcineurin-inhibitor immunosuppressant, is available for oral administration as extended-release tablets containing the equivalent of 0.75 mg, 1 mg, or 4 mg of anhydrous tacrolimus USP. Inactive ingredients include hypromellose USP, lactose monohydrate NF, polyethylene glycol NF, poloxamer NF, magnesium stearate NF, tartaric acid NF, butylated hydroxytoluene NF, and dimethicone NF. Tacrolimus is the active ingredient in ENVARSUS XR.
  Dosage was clinically determined, dose form was oral tablets, and experimental envarsus was once daily
Period: Overall Study
Arm/Group | Standard of Care | Experimental
Started | 50 | 50
Completed | 50 | 48
Not Completed | 0 | 2
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: Tacrolimus (generic; immediate release) is FDA approved for the prophylaxis of organ rejection in heart, kidney and liver transplant recipients.
- Experimental: Envarsus XR is FDA approved for the prophylaxis of organ rejection in kidney transplant recipients converted from tacrolimus immediate-release formulations, in combination with other immunosuppressants. Envarsus XR, is designed to deliver tacrolimus more smoothly over the whole day.
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Experimental | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 5 | 5 | 10
  40-49 years | 8 | 11 | 19
  50-59 years | 21 | 10 | 31
  60-69 years | 12 | 17 | 29
  70-79 years | 4 | 7 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 31 | 38 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 47 | 45 | 92
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 15 | 30
  White | 29 | 32 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Needed to Recover From Delayed Graft Function (DGF)
Description: The primary endpoint of the study will be the length of time between first dialysis and last dialysis after kidney transplant (duration of DGF).
Time Frame: up to 3 months post transplant
Population: 2 patients in SOC and 1 patient in Experimental groups were excluded in analysis due to patients having primary nonfunction of the graft
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care | Experimental
Number analyzed (Participants) | 48 | 49
days | 14.0 [7.5 to 21.0] | 15.0 [9.0 to 20.0]

2. Secondary Outcome: Number of Tacrolimus or Envarsus XR Dose Adjustments Required During the Period of DGF
Description: The secondary endpoint will be number of tacrolimus or Envarsus XR dose adjustments required during the period of DGF.
Time Frame: up to 3 months post transplant
Measure: Median (Inter-Quartile Range); unit: dose adjustments
Arm/Group | Standard of Care | Experimental
Number analyzed (Participants) | 48 | 49
dose adjustments | 4.0 [3.0 to 6.0] | 3.0 [2.0 to 5.0]

3. Other Pre Specified Outcome: Number of Participants Experiencing Related Adverse Events
Description: Number of participants having adverse event will be reported. Adverse events includes the events such as: infections, malignancies, hematological complications including leukopenia, anemia, and thrombocytopenia, cardiovascular complications and events, neuropathy, tremors, gastrointestinal symptoms, uncontrolled hypertension, serious electrolytes abnormalities and immunosuppression-related adverse effects.
Time Frame: up to 3 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Experimental
Number analyzed (Participants) | 50 | 50
Participants | 50 | 48

ADVERSE EVENTS:
Time Frame: up to 3 months
Description: The occurrence of an Adverse Event or Serious Adverse Event may come to the attention of study personnel during study visits and interviews of a study participant presenting for medical care, or upon review by a study monitor.
Arm/Group | Standard of Care | Experimental
All-Cause Mortality (participants affected / at risk) | 0/50 | 2/50
Serious Adverse Events (participants affected / at risk) | 23/50 | 26/50
Other Adverse Events (participants affected / at risk) | 50/50 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=50) | Experimental (N=50)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Other (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 3 (4) | 1 (1)
Other (Cardiac disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2)
Other (Gastrointestinal disorders) | 4 (4) | 3 (3)
Edema (General disorders) | 0 (0) | 1 (1)
Other (General disorders) | 0 (0) | 4 (4)
Common bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
C.Difficile (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Surgical Site Infection (Infections and infestations) | 2 (2) | 0 (0)
Infections and Infestations - Other (Infections and infestations) | 5 (6) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Incisional dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Other (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other (Nervous system disorders) | 0 (0) | 1 (3)
fluid collection around kidney transplant (Surgical and medical procedures) | 6 (6) | 5 (5)
Hydronephrosis (Renal and urinary disorders) | 1 (2) | 0 (0)
Other (Renal and urinary disorders) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Other (Vascular disorders) | 2 (3) | 1 (1)
Hematoma (Vascular disorders) | 2 (2) | 6 (6)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=50) | Experimental (N=50)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Other (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 3 (4) | 2 (2)
Other (Cardiac disorders) | 1 (1) | 2 (2)
visual changes (Eye disorders) | 1 (1) | 0 (0)
Other (Eye disorders) | 1 (1) | 0 (0)
Secondary hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 37 (48) | 28 (44)
Acid Reflux (Gastrointestinal disorders) | 9 (9) | 2 (2)
Nausea (Gastrointestinal disorders) | 14 (14) | 18 (23)
Vomiting (Gastrointestinal disorders) | 11 (13) | 6 (9)
Other (Gastrointestinal disorders) | 6 (8) | 6 (6)
Chills (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (2)
Edema (General disorders) | 10 (11) | 13 (14)
Other (General disorders) | 3 (3) | 5 (5)
Common bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
C.Difficile (Infections and infestations) | 2 (2) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 5 (5)
Surgical Site Infection (Infections and infestations) | 2 (2) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 3 (3)
Infections and Infestations - Other (Infections and infestations) | 6 (7) | 7 (7)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1)
Incisional dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 3 (4)
Other (Injury, poisoning and procedural complications) | 1 (1) | 9 (10)
Weight increase of 5lb in 1 week (Investigations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Other (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Other (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 9 (10) | 5 (7)
Hand tremor (Nervous system disorders) | 22 (25) | 26 (28)
Headache (Nervous system disorders) | 9 (12) | 11 (14)
Other (Nervous system disorders) | 3 (3) | 3 (6)
fluid collection around kidney transplant (Surgical and medical procedures) | 6 (6) | 6 (6)
Hematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (2) | 1 (1)
Other (Renal and urinary disorders) | 6 (6) | 7 (7)
Scrotal Edema (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Other (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Other (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Other (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Other (Vascular disorders) | 2 (3) | 1 (1)
Hematoma (Vascular disorders) | 3 (3) | 6 (6)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT03864926/Prot_SAP_000.pdf